CLINICAL TRIAL: NCT02387567
Title: Study on the Effects of Paraspinal Lidocaine Injection on Nonspecific Low Back Pain
Brief Title: Paraspinal Block in Nonspecific Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marta Imamura (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Sponsor-Investigator, Marta Imamura, 1. Head of Technical Section of Physical and Rehabilitation Medicine of the Orthopedics and Traumatology Institute of HC FMUSP, Coordinator of the Center for Physical and Rehabilitation Medicine of HC FMUSP, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS-block-Pain; U1111-1155-7609 (Other: WHO-UTN U1111-1155-7609)
Record Dates: First submitted 2014-05-22; First posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Lidocaine; Injections; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lidocaine (Experimental): Paraspinal infusion of 3ml lidocaine at 1%, once a week for three weeks, combined with standard treatment.
  Interventions: Drug: Lidocaine; Other: Standard treatment
- Sham lidocaine (Sham Comparator): Sham Injection, without lidocaine, combined with standard treatment.
  Interventions: Drug: Sham Lidocaine; Other: Standard treatment
- Standard treatment only (Active Comparator): The only intervention is the standard treatment. No lidocaine or shame injection was used.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Drug: Lidocaine — Paraspinal block with 3ml lidocaine injection at 1%.
  Other Names: 3ml lidocaine 1% Injection
  Arms: Lidocaine
Drug: Sham Lidocaine — Sham injection, without lidocaine.
  Other Names: 3ml sham injection
  Arms: Sham lidocaine
Other: Standard treatment — Standard treatment only, without lidocaine or sham injection.
  Other Names: Lowback pain standard treatment

SUMMARY:
The purpose of this study is to investigate the effects of a treatment involving the application of lidocaine injected on the low back area for pain control. The study will compare this form of treatment with other options such as physical exercises or pain killer medication, different measurements are going to be used to quantify the response to each of these treatments.

DETAILED DESCRIPTION:
This trial was conducted in the Department of Rehabilitation, Hospital das Clinicas, University, of Sao Paulo Medical School, one of the largest rehabilitation centers in Brazil. The trial was initiated in January of 2007 and close to enrollment in January of 2013. Investigators included patients with a diagnosis of chronic nonspecific low back pain who were referred from various clinics in São Paulo that were linked to this rehabilitation center. Thus, patients were referred primarily by physiatrists, general practitioners, neurologists, orthopedic surgeons, and physiotherapists.

Participants were randomized to receive: (i) paraspinal lidocaine injection (LID-INJ) and standard treatment, (ii) sham lidocaine injection (SH-INJ) and standard treatment, or (iii) standard treatment only (STD-TTR). Randomization was performed using a computerized random number generator.

Assessments The evaluations were performed by an independent and blinded appraiser before treatment, after 1 week, and 3 months after the end of the applications. Baseline assessments consisted of a demographic and baseline clinical assessment [gender, age, occupation, duration of pain (months), pain intensity, associated diseases, and usual occupation] and a physical examination [measurements of weight and height to calculate body mass index (BMI)].

Primary Outcome Measure The primary outcome measure was the visual analog scale (VAS) score for pain. The VAS comprised a 10-cm ruler from 0 to 10, with 0 corresponding to no pain and 10 corresponding to maximum pain. Patients were asked to rate their average pain in the preceding 24 hs.

Secondary Outcome Measures Investigators also measured low back pain using the Brazilian Roland-Morris tool, which consisted of a specific questionnaire to assess function in patients with low back pain and has been validated in Brazil. Scores range from 0 to 24, wherein higher scores reflect greater disability due to low back pain.

ELIGIBILITY:
Inclusion criteria:

* Age between 20 to 60 years;
* Clinical symptoms of vertebral pain that is unresponsive to symptomatic treatment with anti-inflammatory drugs for 3 months;
* Moderate to severe pain: visual analog scale (VAS) > 4;
* Diagnosis of chronic nonspecific low back pain;
* MiniMental test (MEEM) between 24 and 30;
* Availability to comply with the visits;
* Agree with signing the Informed Consent Form

Exclusion criteria:

* Severe psychiatric disease that requires psychiatric care;
* Neurological disorders (lumbosciatic pain);
* Concurrent fibromyalgia, per the 1990 diagnostic criteria of the American Academy of Rheumatology
* Concurrent rheumatic disease
* History of allergy to lidocaine (used for paraspinal blocks)
* Labor problems
* History of surgery on the lumbar spine
* No availability to visit the clinic for treatment and evaluations.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 378 (Actual)
Dates: Start 2007-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the visual analog scale (VAS) score for pain at week 1 | Baseline, week 1

SECONDARY OUTCOMES:
Change from baseline in pain on the Brazilian Roland-Morris tool at week 1 | Baseline, week 1
Change from baseline in pain on the Brazilian Roland-Morris tool at week 12 | baseline, week 12
Change from baseline in pain on the visual analog scale (VAS) score for pain | Baseline, week 12

OTHER OUTCOMES:
Adverse effects questionnaire | Immediately after intervention and 3 months post application

CONTACTS AND LOCATIONS:
Overall Officials: Marta Imamura, MD, Principal Investigator — Instituto de Medicina Física e Reabilitação HCFMUSP
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Imamura M, Imamura ST, Targino RA, Morales-Quezada L, Onoda Tomikawa LC, Onoda Tomikawa LG, Alfieri FM, Filippo TR, da Rocha ID, Neto RB, Fregni F, Battistella LR. Paraspinous Lidocaine Injection for Chronic Nonspecific Low Back Pain: A Randomized Controlled Clinical Trial. J Pain. 2016 May;17(5):569-76. doi: 10.1016/j.jpain.2016.01.469. Epub 2016 Jan 30. PMID 26828801